CLINICAL TRIAL: NCT06932237
Title: Immune-mediated Pathogenic Mechanisms of Neuro-PASC in Veterans
Acronym: PASC
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: James H. Quillen Department of Veterans Affairs Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: MHBC-006-23S; I01CX002668 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Neuro-PASC; Long COVID
Keywords: COVID-19; Veterans; Cognitive; Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neuro-PASC: All participants enrolled in the study will attend 4 study visits: 1) Screening, 2) Baseline, 3) 6-Month Follow-up, and 4) 12-Month Follow-up. At the Baseline, 6-Month, and 12-Month follow-up, participants will complete an online neuropsychological assessment, questionnaires, blood draw, and saliva collection
- Neuro-PASC-imaging: A subset (60) of Portland VA only participants will be provided with the opportunity to complete an MRI visit at baseline and the 12-month follow-up.

SUMMARY:
Mental health symptoms, including cognitive impairment ("brain fog"), following COVID-19 are of great concern to Veterans. The investigators' research seeks to advance understanding of the long-term effects of COVID-19 on neuropsychiatric and neurological functions, identifying clinically relevant biomarkers and directions for developing and testing therapeutic interventions. To accomplish these objectives the investigators are conducting a longitudinal study at two VA medical centers to: 1) assess and monitor cognitive function and psychiatric symptoms in Veterans post-COVID; 2) evaluate biomarkers of inflammation and signaling pathways associated with viral infection and neuropsychiatric function; and 3) integrate neuropsychiatric and neurological findings with biological data to identify biomarkers and clinical endpoints associated with disease progression or severity, as well as those for promoting brain repair and attenuating those symptoms.

DETAILED DESCRIPTION:
The goal of this research project is to identify the neuroinflammatory mechanisms contributing to post-COVID cognitive deficits and neuropsychiatric symptoms [neuro-PASC (post-acute sequelae of SARS CoV-2 infection)]. This collaborative research effort will also characterize new or worsened mental health symptoms and genetic and environmental risk factors for the incidence and severity of post-COVID neuropsychiatric impairments. Aim 1 will monitor and evaluate cognitive injury and neuro-PASC symptoms and determine whether APOE genotype modulates severity of the cognitive injury and neuro-PASC symptoms. Cognitive functioning will be evaluated over time using neuropsychological measures assessing domains most relevant to PASC: learning and memory, attention/concentration, social cognition/emotions, and executive function; assessments will include standardized measures. Mental health symptoms known to be induced and exacerbated by inflammation and potentially developing as a result of COVID-19 will also be evaluated. APOE genotyping will be determined based on saliva or blood samples. Aim 2 will identify immune-related biomarkers associated with cognitive injury and neuro-PASC symptoms. Blood (plasma and cells) will be used to identify biomarkers associated with PASC progression or severity, promotion of brain repair, attenuation of symptoms. Plasma will be used for Olink proteomics, followed by confirmatory multiplex assays or enzyme-linked immunosorbent assays (ELISAs). The investigators will assess relationships among biomarkers and cognitive injury and neuro-PASC symptoms across APOE genotypes and contribute data and samples to the repository managed by Dr. Moorman (Co-Investigator). Aim 3 (exploratory aim; conducted in Portland only) will assess neuroimaging correlates of cognitive injury and neuro-PASC symptoms. Neuroimaging evaluations (i.e., whole brain voxel-based morphometry, diffusion-tensor imaging, resting-state connectivity, and task-based assessments) will be conducted at baseline and at 12 months to correlate magnetic resonance imaging (MRI) measures with symptoms of long COVID (e.g., cognitive impairment and neuropsychiatric symptoms) across APOE genotypes.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will:

* have a history of SARS-CoV-2 infection 4 weeks prior to enrollment, defined as a positive PCR or home antigen test
* be able to give informed consent as determined by brief cognitive exam and evaluation of understanding of the risks, benefits, and voluntary nature of the study

Additionally, participants enrolled as part of the neuro-PASC group must also:

* currently experience neuro-PASC symptoms, not present prior to infection, as confirmed by the "Long COVID-19 Symptom Assessment" scale, a self-report measure that consists of 46 common COVID-19 sequela symptoms

Exclusion Criteria:

Exclusion criteria for all groups:

* diagnosed with dementia, traumatic brain injury, a neurological syndrome (e.g. Parkinson disease, Alzheimer disease), or other progressive cognitive disorder before SARS-CoV-2 infection
* diagnosed with a mood or psychotic disorder before SARS-CoV-2 infection
* history of fibromyalgia or chronic fatigue syndrome prior to SARS-CoV-2 infection
* unstable medical conditions or active uncontrolled autoimmune or inflammatory conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline, 6-Month, 12-Month
  A nine-item self-report questionnaire designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders.
Prospective and Retrospective Memory Questionnaire (PRMQ) | Baseline, 6-Month, 12-Month
  A self-report measure of everyday memory, assessing prospective (the ability to remember to do things in the future) and retrospective memory.
Spatial Working Memory (SWM) | Baseline, 6-Months, 12-Months
  Online cognitive assessment requiring retention and manipulation of visuospatial information; measures executive functioning (i.e., strategy) and working memory.
Paired Associates Learning (PAL) | Baseline, 6-Month, 12-Month
  Online cognitive assessment measuring visual memory and new learning.
Stockings of Cambridge (SOC) | Baseline, 6-Month, 12-Month
  Online cognitive assessment measuring problem-solving strategies.
Delayed Matching Sample (DMS) | Baseline, 6-Month, 12-Month
  Online cognitive assessment measuring visual matching ability and short-term visual recognition memory.
Rapid Visual Information Processing (RVP) | Baseline, 6-Month, 12-Month
  Online cognitive assessment measuring sustained attention.
Apolipoprotein E (APOE) Genotyping | Baseline, 6-Months, 12-Months
  A genetic test that determines a person's inherited variations in the APOE gene. This gene plays a role in cholesterol metabolism and brain health. Blood and saliva samples will be used.
Long Covid Questionnaire | Baseline
  Self-report measure that assesses the continued presence of Long-COVID symptomology.
Delis-Kaplan Executive Functioning - Verbal Fluency (D-KEFS-VF) | Baseline, 6-Months, 12-Months
  Neuropsychological assessment measure of verbal behavioral productivity and cognitive flexibility.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist - Civilian Version (PCL-C) | Baseline, 6-Month, 12-Month
  A standardized self-report rating scale for PTSD comprising 17 items that correspond to the key symptoms of PTSD.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 6-Months, 12-Months
  Self-report questionnaire objectifying and assessing degree of depression severity.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 6-Month, 12-Month
  A self-reported questionnaire used to assess the severity of anxiety symptoms.
Biomarkers | Baseline, 6-Months, 12-Months
  Obtained from collected blood samples and saliva, biomarkers (including viral variants, genetic susceptibility, inflammatory markers, diagnostic markers, etc.) associated with specific symptoms of post-COVID conditions will be identified.

OTHER OUTCOMES:
Neuroimaging | Baseline, 12-Months
  To detect pathological and restorative changes in the brain of COVID-19 survivors, neuroimaging evaluations will correlate magnetic resonance imaging (MRI) measures with symptoms of neuro-PASC.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Loftis, MA PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (2):
- United States (2):
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee

IPD SHARING:
Plan to Share IPD: No